CLINICAL TRIAL: NCT07269548
Title: Evaluation of the Healing of the Pilonidal Cyst After 1940 nm Laser Treatment
Acronym: PILOLAS 1940
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-06-045-P-ERAMD0619
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pilonidal Cyst/Fistula
Keywords: healing, Pilonidal Cyst
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LASER 1940: Patient who underwent surgery for a pilonidal cyst using 1940 nm laser treatment
  Interventions: Procedure: pilonidal cyst laser surgery

INTERVENTIONS:
Procedure: pilonidal cyst laser surgery — pilonidal cyst using 1940 nm laser treatment

SUMMARY:
The aim of this study is to evaluate the extent to which the reduction of energy absorption that laser 1940 nm allows could improve the outcomes and postoperative results of the treatment of pilonidal cysts.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not object to the collection of their data
* Patients who underwent surgery for a pilonidal cyst using 1940 nm laser treatment

Exclusion Criteria:

* Patients with a history of pilonidal cyst surgery

  * Patients who underwent emergency surgery for an abscess
  * Patients already included in another therapeutic study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with laser 1940 nm for a pilonidal cyst.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HEALING | 1 Month
  The main objective is to evaluate the healing rate of the pilonidal sinus one month after treatment with Er-YAG laser 1940 nm. Wound healing at one month, defined by the absence of a dressing, is the main evaluation criterion.

SECONDARY OUTCOMES:
Recidivism | 6 Month
  Recidivism is defined by: - The presence of persistent troubling symptoms 6 months after the surgery: suppuration, recurrent wound dehiscence, lack of healing despite care deemed optimal by the expert, reactivation/recurrence of abscesses. - The presence of a characteristic image on MRI if this examination has been carried out: subcutaneous collection, in hyper T2.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France